CLINICAL TRIAL: NCT01128361
Title: Alzheimer's Disease Exercise Prevention Trial
Brief Title: Pilot Study of Aerobic Exercise in Early Alzheimer's Disease(AD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeff Burns, MD (Other)
Responsible Party: Sponsor-Investigator, Jeff Burns, MD, Assistant Professor, Director of the Alzheimer & Memory Center & AD Clinical Research Program, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11969
Record Dates: First submitted 2010-05-18; First posted 2010-05-21 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic Exercise (Experimental)
  Interventions: Behavioral: Aerobic Exercise
- Stretching (Active Comparator)
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Aerobic Exercise — Participants randomized to this group will perform 150 minutes a week of aerobic exercise over 3-5days. Participants will begin exercising 3 times the first week for 20 minutes, increasing to three bouts of 25 minutes the second week. Thereafter, weekly exercise duration will be increased until their target duration of 150 minutes is achieved in week 6. Exercise trainers will assist participants in adjusting exercise routines to achieve their weekly exercise duration goals. Use of equipment, achievement of target HR and safety will be closely monitored by the trainer through the course of the study. Each subject will wear a Polar F4 heart monitor (Polar USA) for recording heart rate during each exercise session. Subjects unable to exercise continuously on the treadmill will perform intermittent training until the target duration is reached. The majority of the exercise sessions will involve walking on a treadmill.
  Arms: Aerobic Exercise
Behavioral: Stretching — This groups intervention is designed to match the aerobic exercise intervention with respect to participation and socialization. Stretching and toning has been repeatedly used as control intervention for exercise studies.The schedule and format will be identical to the aerobic conditioning group to best balance confounding variables such as attention, social interactions, and other unknown variables that might influence the results. An experienced and trained exercise instructor will run the stretching sessions three days a week at the local YMCA. We will monitor changes in heart rate with Polar F4 heart monitors (Polar USA) during the sessions to assess, and minimize, potential aerobic benefits from the intervention.
  Arms: Stretching

SUMMARY:
The current project is a natural extension of a programmatic line of investigation into the relationship between exercise, brain aging, and AD that Dr. Burns has developed over the last four years. The current study will provide data to estimate expected effect sizes for power analyses and sample size calculations. It will also provide an opportunity to optimally design a larger trial that can be extended to multiple sites to more definitively examine the role of exercise as a therapy in AD. The current project's aims are an important and necessary developmental step given the lack of fitness data in AD and the limited knowledge of the mechanisms that may form the basis of an association between aerobic fitness and AD.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided by the participant or the participant's legally acceptable representative
* Age 55 years or older
* Diagnosis of Probable AD according to the National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA)
* Clinical Dementia Rating (CDR) of 0.5 (very mild) or 1 (mild dementia)
* Mini-Mental Status Exam Score of 16 to 30, inclusive.
* Rosen Modified Hachinski score of 4 or less
* Community dwelling with a caregiver able and willing to accompany the participant on all visits, if necessary. The caregiver must visit with the subject more than five times a week for the duration of the study.
* Underactive or sedentary as determined by a Telephone Assessment of Physical Activity.
* Adequate visual and auditory abilities to perform all aspects of the cognitive and functional assessments
* Stable doses of medications for at least 30 days prior to screening. Cholinesterase inhibitors and memantine are allowed provided the participant is on stable doses without clinically significant side effects for 60 days. Additionally, the participant and caregiver will agree, barring unforeseen circumstances, to continue the same regimen for the trial duration.
* Likely to participate in all scheduled evaluations and complete the 26 week program.

Exclusion Criteria:

* CDR 0.5 uncertain dementia (i.e., not meeting NINCDS-ADRDA criteria).
* Significant neurological disease, other than AD, that may affect cognition
* MRI or CT scan indicative of significant abnormalities that may explain cognitive decline (e.g., multiple lacunar infarcts or a single prior infarct > 1 cm3, micro-hemorrhages or evidence of a prior hemorrhage > 1 cm3, evidence of cerebral contusion, encephalomalacia, aneurysm, vascular malformation, or space-occupying lesion such as an arachnoid cyst or brain tumor)
* Current clinically significant major psychiatric disorder (e.g., Major Depressive Disorder) according to DSM-IV criteria or significant psychiatric symptoms (e.g., hallucinations) that could impair the completion of the study. Individuals with depressive symptoms (Geriatric Depression Scale < 6) and who do not meet criteria for major depression will be eligible.
* Current clinically-significant systemic illness that is likely to result in deterioration of the patient's condition or affect the patient's safety during the study
* History of clinically-evident stroke
* Clinically-significant infection within the last 30 days
* Myocardial infarction or symptoms of coronary artery disease (e.g., angina) in the last two-years.
* Uncontrolled hypertension within the last 6 months
* History of cancer within the last 5 years (except non-metastatic basal or squamous cell carcinoma)
* History of drug or alcohol abuse as defined by DSM-IV criteria within the last 2 years
* Presence of contraindications for MRI scanning (pacemaker, aneurysm clips, artificial heart valves, metal fragments, foreign objects) or claustrophobia
* Insulin-dependent diabetes mellitus
* Significant pain or musculoskeletal disorder that would prohibit participation in an exercise program

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Burns, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Morris JK, Vidoni ED, Johnson DK, Van Sciver A, Mahnken JD, Honea RA, Wilkins HM, Brooks WM, Billinger SA, Swerdlow RH, Burns JM. Aerobic exercise for Alzheimer's disease: A randomized controlled pilot trial. PLoS One. 2017 Feb 10;12(2):e0170547. doi: 10.1371/journal.pone.0170547. eCollection 2017. PMID 28187125

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aerobic Exercise | Stretching
Started | 39 | 37
Completed | 34 | 34
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise | Stretching | Total
Number analyzed (Participants) | 39 | 37 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 39 | 37 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.4 (6.7) | 71.4 (8.4) | 72.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 21 | 16 | 37
Region of Enrollment [Number; unit: participants]
  United States | 39 | 37 | 76
Clinical Dementia Rating Sum of Boxes [Mean (Standard Deviation); unit: units on a scale] — The Clinical Dementia Rating (CDR) is a scale used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care. The sum of each domain (CDR Sum of Boxes) is used as a measure of dementia severity from 0 (no impairment) to 18 (severe impairment).
  units on a scale | 3.54 (1.99) | 3.55 (1.60) | 3.54 (1.81)

OUTCOME MEASURES:

1. Primary Outcome: Memory Composite
Description: A composite measure of several memory tests (Logical Memory (Immediate and Delayed), Free and Cued Selective Reminding Test (sum of free recall). Each score was normalized to an independent dataset of individuals without dementia. Then the 4 standardized scores were averaged.
  Numbers closer to positive indicate better memory performance. The scores are centered around a mean of 0 and standardized so each value represents a fraction of the standard deviation. There are no limits to the scores.
Time Frame: week 0, 13, and 26
Population: Linear mixed models with all available data were used. Thus the overall number of participants analyzed does not necessarily match the means reported at each timepoint.
Measure: Mean (Standard Deviation); unit: units on a standardized scale
Arm/Group | Aerobic Exercise | Stretching
Number analyzed (Participants) | 39 | 37
units on a standardized scale
  Baseline | -2.5 (1.4) | -2.8 (1.4)
  Week 13: number analyzed (Participants) | 36 | 37
  Week 13 | -2.3 (1.5) | -2.8 (1.5)
  Week 26: number analyzed (Participants) | 34 | 34
  Week 26 | -2.3 (1.7) | -2.7 (1.7)

2. Primary Outcome: Executive Function Composite
Description: A composite measure of several memory tests (Logical Memory (Immediate and Delayed), Free and Cued Selective Reminding Test (sum of free recall). Each score was normalized to an independent dataset. Then the 4 standardized scores were averaged.
  Numbers closer to positive indicate better executive function performance. . The scores are centered around a mean of 0 and standardized so each value represents a fraction of the standard deviation. There are no limits to the scores.
Time Frame: Week 0, 13, and 26
Population: Linear mixed models were used with all available data included. Overall numbers analyzed do not necessarily match the outcome measure at each timepoint
Measure: Mean (Standard Deviation); unit: standardized units on a scale
Arm/Group | Aerobic Exercise | Stretching
Number analyzed (Participants) | 39 | 37
standardized units on a scale
  Baseline | -1.12 (.82) | -1.34 (.85)
  Week 13: number analyzed (Participants) | 36 | 37
  Week 13 | -1.09 (.86) | -1.25 (.94)
  Week 26: number analyzed (Participants) | 34 | 34
  Week 26 | -1.2 (.9) | -1.33 (.97)

3. Primary Outcome: Disability Assessment for Dementia
Description: This is a validated measure of disability for individuals with dementia. Higher scores indicate less disability with a score of 100 indicating no disability and 0 indicating no functional ability.
Time Frame: Week 0, 13, and 26
Population: Linear mixed models were used with all available data. Overall number of participants may not match numbers at each timepoint.
Measure: Mean (Standard Deviation); unit: percentage on a scale
Arm/Group | Aerobic Exercise | Stretching
Number analyzed (Participants) | 39 | 37
percentage on a scale
  Baseline | 88 (12.3) | 91.2 (8)
  Week 13: number analyzed (Participants) | 36 | 37
  Week 13 | 89.8 (12.5) | 89.5 (12.8)
  Week 26: number analyzed (Participants) | 34 | 34
  Week 26 | 89.5 (13.7) | 86.7 (13.3)

4. Primary Outcome: Cornell Scale for Depression in Dementia
Description: The Cornell Scale for Depression in Dementia is a validate measure of depressive symptoms in individuals with dementia. Larger numbers indicate greater levels of depression. Scores range from 0 to 38.
Time Frame: Week 0, 13, and 26
Population: Linear mixed models were used with all available data. Overall numbers analyzed may not reflect numbers at each timepoint
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise | Stretching
Number analyzed (Participants) | 39 | 37
units on a scale
  Baseline | 7.4 (3.8) | 8.6 (5.1)
  Week 13: number analyzed (Participants) | 36 | 37
  Week 13 | 8.1 (4.4) | 8.4 (4.6)
  Week 26: number analyzed (Participants) | 34 | 34
  Week 26 | 7.8 (4.4) | 7.8 (5.2)

ADVERSE EVENTS:
Arm/Group | Aerobic Exercise | Stretching
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/37
Other Adverse Events (participants affected / at risk) | 13/39 | 9/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise (N=39) | Stretching (N=37)
Cardiac (Cardiac disorders) | 8 (8) | 4 (4) — Arrhythmia or EKG abnormality noted on exercise testing
Muscle soreness or joint pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin breakdown (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No